CLINICAL TRIAL: NCT01230359
Title: EARLY NUTRITIONAL INTERVENTION IN PATIENTS WITH AUTISM SPECTRUM DISORDERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Qatar University (Other); Heidelberg University (Other)
Responsible Party: Dr. Fadhila Al -Rawi, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8225/08
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Autism Spectrum Disorders; Stable Clinical Condition in the Last 3 Months
Keywords: Autism; Children; ASD; Vitamin B6; Magnesium
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Pyridoxine; Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin B6 and magnesium (Experimental)
  Interventions: Dietary Supplement: Pyridoxine hydrochloride
- Tang powder group (Placebo Comparator)
  Interventions: Other: Tang orange powder

INTERVENTIONS:
Dietary Supplement: Pyridoxine hydrochloride — 2.5 grams per day for subjects weighing upto 27 kilos and 5 g per day for greater than 27 kgs for 12 weeks
  Other Names: Vitamin B6; Super Nu -Thera Registered trade mark kirkman Laboratories
  Arms: Vitamin B6 and magnesium
Other: Tang orange powder — 2.5 grams per day for subjects weighing upto 27 kilos and 5 g per day for greater than 27 kgs for 12 weeks
  Arms: Tang powder group

SUMMARY:
Nutritional supplements like vitamin B6 and magnesium have demonstrated to have beneficial effects in patients with autism spectrum disorders (ASD). The underlying theory for these effects is that specific metabolic pathways in neuronal cells, e.g. the methionine cycle, will be more balanced. Most studies have been focused on the clinical outcome with this treatment. The present proposal will examine the effects on the different intermediates of the methionine cycle (methylation and transulfuration capacity), suggested to play an important role for the pathogenesis of ASD. The design is a prospective pilot study, including 40 patients, aged 2-6 yrs, with newly diagnosed ASD. All participants will receive the supplement (vitamin B6, magnesium; Kirkman formula) and placebo in a cross over design. Metabolites in blood and urine will be measured prior to and at the end of the treatments in the different groups. The results will then provide us with information, which will link clinical outcomes with biological markers. Furthermore, the study has also the potential to shed light on the pathogenesis of ASD.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASDs) are neurodevelopment disorders characterized by impairments in social relatedness and communication, repetitive behaviors, abnormal movement patterns, and sensory dysfunction that affect children from birth or the early months of life, but only recognized by most parents between 12 and 24 months of age.

Studies have shown that a diagnosis of autism can be reliably made between 2 and 3 years of age, although a diagnosis of the broader autistic spectrum is less reliable at this age than in older children While genetic factors are recognized as being important in the pathogenesis of ASDs, a metabolic and biochemical factors are considered to play an important role for the pathogenesis. Treatment is directed on the impairing core features of the disorder.

Pyridoxine (vitamin B6) was first used with children diagnosed with "autism syndrome" when speech and language improvement was observed in some children as a result of large doses of B6. Magnesium was added to prevent the possibility of hyperactivity and peripheral neuropathy, which can occur if the vitamin B6 is taken by itself. An impairment of the methionine cycle and transsulfuration was previously reported in autistic children. Recent studies in autistic children have suggested a decreased capacity for methylation as contributing factor to the development and clinical manifestation of the disease .

Homocysteine is removed either by its irreversible conversion to cysteine (transsulfuration) or by remethylation to methionine. There are two separate remethylation reactions, catalyzed by betaine. The reactions that remove homocysteine are very sensitive to B vitamin status as both the transsulfuration enzymes contain pyridoxal phosphate, while methionine synthase contains cobalamin and receives its methyl group from folic acid one-carbon pool.

In addition, vitamin B6 is required for over 100 enzymatic reactions, including the production of major neurotransmitters (serotonin, dopamine, and others) and glutathione (needed for detoxification).

A number of studies attempted to assess the effects of vitamin B6-Magnesium (Mg) on characteristics such as verbal communication, non-verbal communication, interpersonal skills, and physiological function, in individuals with autism. There are over 22 studies of vitamin B6 with Magnesium for ASD, including 11 double-blind, placebo-controlled studies, making it one of most studied treatments for autism. Many of these studies found some of the children with ASD benefited from high-dose supplementation of vitamin B6 with Magnesium in many areas of the spectrum including language, eye contact and behaviour . Twenty-one of these yielded positive results, and only minor adverse effects were reported , In the Cochrane Database Systematic Review only study yielded no significant performances between treatment and placebo group performances following the B6 intervention on measures of social interaction, communication, compulsivity, impulsivity or hyperactivity.

However, none of the above studies evaluated the effect of the vitamin B6 on the methionine cycle.

In summary, the proposed study will compare biochemical alterations in a key metabolic pathway, i.e. the methionine cycle, suggested by previous studies to play an important role in the pathogenesis of ASD, with clinical parameters, during treatment with nutritional supplement. Therefore, the results will provide clinicians with important information for improvement and optimization of the treatment of patients with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2-6 years of age referred to Pediatrics Rehabilitation Clinic with suspected ASD and pre-screened with DSM IV-R.
* Each patient will be free of psychoactive medication for at least 3 months prior to the entry into the trial.

Exclusion Criteria:

* - Patients with chronic illness or known hormonal or metabolic disease.
* Patients with known genetic or chromosomal syndromes.
* Inability of parents to give informed consent, travel to the clinic visits, administer study medication or arrange for completion of rating scales.

We will not to exclude children on other concurrent medications (e.g. antibiotics for intercurrent illnesses, etc.) but will record these medications and control their presence in the final analysis. Furthermore, we will not to exclude children with other co- morbid neurological disorders (e.g. seizure disorder may be present in up to 25% of autistic patients). We will record these conditions and use them in the predictor model to understand their relationship with our current management protocol.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Measurement of improvement in blood parameters | At 12 weeks after getting the nutritional supplement
  Nutritional supplement is provided and the measures of blood tests are done 12 weeks after the participant takes the supplement

SECONDARY OUTCOMES:
Developmental assessments for ASD | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rumailah Hospital, Doha, Qatar, Qatar